CLINICAL TRIAL: NCT04834128
Title: A Phase II Safety and Tolerability, Inter-patient Pre-defined Dose Study of Ex-vivo Expanded Allogeneic γδ T-lymphocytes (TCB008) in Patients Diagnosed With COVID-19
Brief Title: A Phase II Safety and Tolerability Study of TCB008 in Patients With COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped because of the current status of the COVID-19 epidemic in the United Kingdom, and also because the trial involved parenterally administered IMP and a period of inpatient care and extensive outpatient visits and investigations.
Sponsor: TC Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCB008-002
Record Dates: First submitted 2021-03-29; First posted 2021-04-06 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: COVID - 19
Keywords: ATMP
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: open-label, safety and tolerability, escalating dose, single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- γδ T cells (IMP, TCB008) (Experimental): Patients will receive an infusion of γδ T cells (IMP, TCB008) following informed consent after admission to hospital for SARS-CoV-2 infection (COVID-19).
  Interventions: Drug: TCB008

INTERVENTIONS:
Drug: TCB008 — administration of gamma delta T cells by IV bolus injection

SUMMARY:
A Phase II safety and tolerability study of expanded gamma delta T cell lymphocytes (TCB008) in patients diagnosed with COVID-19.

DETAILED DESCRIPTION:
The aim of this Phase II study is to evaluate the safety and tolerability of ex-vivo expanded gamma delta T-cells (TCB008) manufactured from a single allogeneic unmatched or partially, randomly matched, unrelated donor, in patients with COVID-19.

The trial is designed to identify an optimal, safe dose of allogeneic γδ T cells in a population of patients with COVID-19. There will be 4 patient Cohorts. Cohorts 1 - 3 will receive a pre-defined dosing schedule, with Cohort 4 being treated with a dose selected upon completion of the first 3 Cohorts. In order to investigate immunogenicity assessment/sensitisation effects, patients in the expansion cohort who do not experience adverse reactions meeting dose limiting toxicity (DLT) criteria after the first administration will receive re-infusion with the same dose on Day 10 after the first infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participating in the clinical study; fully understanding and being fully informed of the study and having signed the Informed Consent Form (ICF);

   - willingness and capability to complete all the study procedures
2. Age 18-65 years (inclusive) at the time of signing ICF
3. Any gender
4. Patients with a positive diagnosis of COVID-19 either identified in the community as at risk of progression of disease or

   * already hospitalized with new changes on CXR or CT scan compatible with COVID19, or
   * patients requiring supplemental oxygen, but for whom dexamethasone is not yet indicated according to current standard of care recommendations.

The product would be indicated for patients categorized as per the WHO ordinal scale 2,3 or 4: i.e., ambulatory (or community identified) patients with limitations of activity, judged as at risk for progression of disease, as well as hospitalized patients not yet requiring oxygen therapy or receiving non-invasive low flow oxygen therapy, which does not yet indicate the need to commence dexamethasone therapy.

Exclusion Criteria

1. Patients requiring high-flow oxygen therapy and/or dexamethasone according to the current standard of care.
2. Patients suffering from severe cognitive impairment or mental illness
3. Pregnant and/or lactating women
4. Patients participating in other CTIMP clinical studies at the same time
5. Active autoimmune disease or Graft versus Host Disease (GVHD)
6. Patients with any major comorbidity (e.g., diabetes, cardiovascular and pulmonary diseases, malignancies on active treatment) unless their pre-morbid Karnofsky performance status was ≥ 80%
7. Patients with documented history of immunological disorders
8. Immunocompromised patients defined as those with human immunodeficiency virus infection with a CD4 cell count of less than 200 per microliter or uncontrolled viremia, prolonged use of glucocorticoids or other immunomodulating medications, a history of bone marrow or organ transplantation
9. ALT / AST> 5 times the upper limit of the normal
10. Neutrophils <500 / mm3
11. Platelets <50.000 / mm3
12. Patients known or suspected to have sensitivity against mouse immunoglobulins or iron-dextran.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Assessment of treatment emergent adverse events (AEs) - Safety | 30 and 90 days after IMP administration
  Safety of IMP assessed by incidence of treatment-emergent adverse events (AEs) per patient, graded by Common Terminology Criteria for Adverse Events (CTCAE) V5.0
Incidence of dose-limiting toxicities (DLTs) - Tolerability | 30 and 90 days after IMP administration
  Tolerability of IMP assessed by incidence of dose-limiting toxicities (DLT's) graded by Common Terminology Criteria for Adverse Events (CTCAE) V5.0
Establish Maximum Tolerated Dose (MTD) or Maximum Feasible Dose (MFD) - Tolerability | Approx 1 year
  Tolerability of IMP assessed by incidence of dose-limiting toxicities (DLT's) graded by Common Terminology Criteria for Adverse Events (CTCAE) V5.0

OTHER OUTCOMES:
Persistence of gamma delta T cells | Approx 1 year
  Assessment of the persistence of gamma delta T cells in the peripheral blood os dosed patients using flow cytometry
Phenotype of gamma delta T cells | Approx 1 year
  Assessment of the phenotype of gamma delta T cells in the peripheral blood of dosed patients using flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Victoria Infirmary, Newcastle, United Kingdom